CLINICAL TRIAL: NCT07384026
Title: An International Study on the Professional Quality of Life of Youth Care Professionals
Brief Title: International Online Survey Assessing Secondary Traumatic Stress, Burnout, Compassion Satisfaction and Turnover Intentions Among Youth Care (Para)Professionals in Flanders, Wallonia, France and The Netherlands.
Acronym: 2021_VUB_CFCSJ
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universiteit Leiden (Other)
Responsible Party: Sponsor
Other Study IDs: B.U.N. 1432021000667
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Secondary Traumatic Stress; Burnout, Professional; Compassion Fatigue; Compassion Satisfaction; Turnoverintention; Professional Quality of Life
Keywords: Burnout; Secondary Traumatic Stress; Compassion Fatigue; Compassion Satisfaction; Turnover; Child Welfare; Foster Carer
MeSH Terms: conditions — Compassion Fatigue; Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth Care (Para)Professionals: This cohort consists of adults working as (para)professionals in youth care services in Flanders, Wallonia, France and The Netherlands. Participants share the common exposure of providing direct support to children and adolescents who may have experienced trauma. All participants complete a single, anonymous online survey assessing personal, work-related, and client-related factors as well as measures of secondary traumatic stress, burnout, compassion satisfaction, and turnover intention. No intervention is administered, and no follow-up occurs; the cohort represents a single cross-sectional observational group.

SUMMARY:
The goal of this observational study is to understand how work-related stress and personal characteristics affect the wellbeing of adults who work with children and young people in youth care services in Flanders, Wallonia, France and The Netherlands. The study focuses on three aspects of professional wellbeing: secondary traumatic stress, burnout, and compassion satisfaction. These feelings can develop when people regularly support children and families who have experienced trauma. The study also looks at whether these experiences influence participants' intention to leave their job.

The main questions this study aims to answer are:

1. What are the levels of secondary traumatic stress, burnout, and compassion satisfaction among youth care (para)professionals?
2. Which personal, work-related, and client-related factors raise or lower the risk of experiencing these outcomes?
3. How do these wellbeing outcomes relate to participants' intention to leave their job?
4. Do these outcomes differ between regions (Flanders, Wallonia, France, The Netherlands) and between types of youth care roles (professional vs. paraprofessional)?

Participants will complete an anonymous online survey that takes about 15 to 20 minutes. The survey asks about everyday work experiences, personal wellbeing, social support, workload, client characteristics, and professional quality of life. All answers are anonymous, and no identifying information (such as names or IP addresses) is collected.

There is no intervention and no comparison group; this study only collects information to better understand the wellbeing of youth care (para)professionals. The goal is to identify challenges and strengths in the sector and to support future prevention and intervention efforts that promote healthy, sustainable working conditions.

The study includes adults who work directly with children or adolescents in youth care settings, such as residential care workers, family support workers, foster care staff, foster carers and other caregiving professionals. People whose roles involve low likelihood of trauma exposure (such as prevention-focused services) are not included.

Ultimately, this research aims to help youth care organizations better support their workforce, reduce work-related stress, and improve continuity and quality of care for children and families.

DETAILED DESCRIPTION:
This observational study examines the professional quality of life of (para)professionals working in youth care services in Flanders, Wallonia, and France. Youth care providers are frequently exposed to the emotional and psychological impact of working with children and adolescents who have experienced trauma. This exposure may contribute to secondary traumatic stress (STS), burnout, and variations in compassion satisfaction. These factors are collectively conceptualized under the Professional Quality of Life (ProQOL) model. Understanding the levels, predictors, and consequences of these outcomes is essential for safeguarding the wellbeing of the workforce and ensuring continuity and quality of youth care services.

The study uses an anonymous online survey developed in Qualtrics. The survey includes structured modules that assess personal factors (e.g., demographic characteristics, social support, financial strain, personality traits, self-care behaviors), work-related characteristics (e.g., workload, work-family conflict, organizational support, colleague support, job role, caseload, type of service), and client-related factors (e.g., client trauma exposure, case complexity, involvement with crisis cases, perceived overinvolvement with clients). These domains are followed by validated instruments measuring the primary outcomes: secondary traumatic stress, burnout, and compassion satisfaction, derived from the Professional Quality of Life Scale Version 5 (ProQOL-5). Turnover intention is assessed using items adapted from previous research in child welfare settings.

Data collection procedures ensure anonymity and confidentiality. IP tracking in Qualtrics is disabled, and no identifying information is stored. Data are downloaded from Qualtrics into a secure, password-protected SharePoint environment hosted by the Vrije Universiteit Brussel. Only authorized members of the research team have access to the dataset. After the response rate per organization is calculated, the variable identifying the participant's employing organization is deleted to prevent potential re-identification.

The statistical analysis plan includes a combination of descriptive and inferential approaches. Descriptive analyses summarize levels of STS, burnout, and compassion satisfaction across regions. Group comparisons between Flanders, Wallonia, France and The Netherlands are conducted using independent samples t-tests or ANOVA, depending on the number of comparison groups. Predictor analyses include Pearson correlations, t-tests, and ANOVA to identify variables associated with each outcome domain at the exploratory level. Subsequently, separate multiple linear regression models are conducted for burnout, STS, and compassion satisfaction, including predictors that showed relations at p ≤ .10 in preliminary analyses. Turnover intention is examined using hierarchical regression to determine whether STS, burnout, and compassion satisfaction explain additional variance beyond personal, work, and client factors. Differences in outcome levels across types of youth care roles (e.g., residential workers, family support workers, foster care staff) are evaluated using t-tests and ANOVA.

To ensure data quality, the dataset is screened for missing values, outliers, and inconsistencies before analysis. Cases with extensive missingness or extreme outliers may be removed. Analyses are performed in IBM SPSS Statistics version 27. The sample size target of approximately 3,000 participants allows for adequate statistical power to detect differences across subgroups and to estimate multivariable models with sufficient precision.

The study is conducted in accordance with ethical principles outlined in the Declaration of Helsinki and Good Clinical Practice guidelines. Data collection is entirely anonymous, and informed consent is obtained electronically prior to participation. Participants may complete the survey at their convenience, and the survey duration is approximately 15 to 20 minutes.

Given the growing pressure on youth care systems and the increasing demand for services, understanding risk and protective factors that shape professional wellbeing is highly relevant. The findings of this study will contribute to developing prevention strategies, informing organizational support systems, and guiding policy decisions aimed at improving working conditions and reducing staff turnover. The results will be disseminated through scientific publications, master's theses, and a doctoral dissertation. National and regional research teams in Belgium, France, and the Netherlands will publish region-specific analyses as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older).
* Currently working as a (para)professional in youth care services.
* Provides support or guidance to children or adolescents who are followed by a youth care organization in Flanders, Wallonia, France or The Netherlands.
* Able to complete an online survey in Dutch or French.
* Provides informed consent electronically.

Exclusion Criteria:

* Works in a youth care service where exposure to client trauma is unlikely (for example, services focused mainly on prevention).
* Works with children or adolescents who are followed primarily due to a disability, without likelihood of trauma exposure.
* Unable to complete the online survey independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults working as (para)professionals in youth care services in Flanders, Wallonia, France, and The Netherlands. Participants are recruited from organizations that provide support, guidance, or protection to children and adolescents, including residential care facilities, family support services, foster care agencies, and other youth care settings. Recruitment occurs through collaboration with youth care organizations and universities in the participating regions. All participants complete a one-time anonymous online survey.
Sampling Method: Non-Probability Sample
Enrollment: 4214 (Actual)
Dates: Start 2022-02-06 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Secondary Traumatic Stress Score on the Professional Quality of Life Scale (ProQOL-5) | Day 1
  Secondary traumatic stress will be measured using the Secondary Traumatic Stress subscale of the Professional Quality of Life Scale Version 5 (ProQOL-5). The scale produces a summed score ranging from 10 to 50, where higher scores indicate higher levels of secondary traumatic stress resulting from indirect exposure to others' trauma. Participants rate how often work-related experiences occurred in the past 30 days on a 5-point Likert scale.
Burnout Score on the Professional Quality of Life Scale (ProQOL-5) | Day 1
  Burnout will be measured using the Burnout subscale of the Professional Quality of Life Scale Version 5 (ProQOL-5). This subscale yields a total score between 10 and 50, with higher scores reflecting higher levels of work-related emotional and physical exhaustion. Items are rated using a 5-point Likert scale based on the frequency of experiences during the past 30 days.
Compassion Satisfaction Score on the Professional Quality of Life Scale (ProQOL-5) | Day 1
  Compassion satisfaction will be measured using the Compassion Satisfaction subscale of the Professional Quality of Life Scale Version 5 (ProQOL-5). Scores range from 10 to 50, with higher values indicating greater satisfaction and positive feelings derived from helping others in one's professional role. Items are rated on a 5-point Likert scale based on experiences in the past 30 days.

SECONDARY OUTCOMES:
Turnover Intention Score on the Turnover Intention Scale | Day 1
  Turnover intention will be measured using items adapted from validated turnover intention scales used in child welfare research (e.g., Prost & Middleton, 2020). The measure assesses the participant's intention to leave their job or the child welfare field. Items are rated on a Likert scale, and scores are summed to produce a continuous value. Higher scores indicate a stronger intention to leave the profession. The expected score range depends on the number of included items, but higher values consistently reflect greater turnover intention.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Vanderfaeillie, PhD, Study Chair — johan.vanderfaeillie@vub.be
Locations (1):
- Vrije Universiteit Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study collects anonymous survey data through Qualtrics, without any identifying information or the ability to link responses to individuals. As described in the protocol, the data will be used exclusively for the purposes of this study and stored securely on a password-protected SharePoint environment of the VUB. Because the dataset contains anonymous responses and no plan for external IPD sharing was defined in the protocol, IPD cannot be made available.

REFERENCES:
- [Background] Maslach, C., Schaufeli, W., & Leiter, M. (2001). Job burnout. Annual Review of Psychology, 52, 397-422.
- [Background] Verheyden, C., Van Holen, F., West, D. & Vanderfaeillie, J. (2020). Secondary traumatic stress, burnout and compassion satisfaction among Flemish foster care workers during the COVID- 19 lockdown. Developmental Child Welfare, 2(4), 227-243. https://doi.org/10.1177/2516103220987227
- [Background] Schaufeli, W.B. & Bakker A.B. (2007). Burnout en bevlogenheid [Burnout and work engagement]. In W.B. Schaufeli & A.B. Bakker (Red.). De psychologie van arbeid en gezondheid (pp. 341- 358). Bohn Stafleu van Loghum.
- [Background] Salloum, A., Kondrat, D. C., Johnco, C. & Olson, K. R. (2015). The role of self-care on compassion satisfaction, burnout and secondary trauma among child welfare workers. Children and Youth Services Review, 49, 54-61. https://doi.org/10.1016/j.childyouth.2014.12.023
- [Background] Mor Barak, M. E., Levin, A., Nissly, J. A. & Lane, C. J. (2006). Why do they leave? Modeling child welfare workers' turnover intentions. Children and Youth Services Review, 28(5), 548-577. https://doi.org/10.1016/j.childyouth.2005.06.003
- [Background] Middleton, J. S. & Potter, C. C. (2015). Relationship Between Vicarious Traumatization and Turnover Among Child Welfare Professionals. Journal of Public Child Welfare, 9(2), 195- 216. https://doi.org/10.1080/15548732.2015.1021987
- [Background] Lizano, E., & Mor Barak, M. (2012). Workplace demands and resources as antecedents of job burnout among public child welfare workers: A longitudinal study. Children and Youth Services Review, 34(9),1769-1776.
- [Background] Gosling, S., Rentfrow, P., & Swann, W. (2003). A very brief measure of the Big-Five personality domains. Journal of Research in Personality, 37(6), 504-528.
- [Background] Figley, C. (1995). Compassion fatigue as secondary traumatic stress disorder: An overview. In C. Figley (Ed.), Compassion fatigue: Coping with secondary traumatic stress disorder in those who treat the traumatized (pp. 1-20). Routledge.
- [Background] Elo, A.-L., Dallner, M., Gamberale, F., Hottinen, V., Knardahl, S., Lindström, K., Skogstad, A., & Ørhede, E. (2000). Validation of the Nordic Questionnaire for Psychological and Social Factors at Work-QPSNordic. In M. Vartiainen, F. Avallone, & N. Anderson (Eds.), Innovative theories, tools, and practices in work and organizational psychology (pp. 47-57). Hogrefe & Huber Publishers.
- [Background] Cornille, T. A. & Meyers, T. W. (1999). Secondary traumatic stress among child protective service workers: Prevalence, severity and predictive factors. Traumatology, 5(1). https://doi.org/10.1177/153476569900500105
- [Background] Chen, Y. Y., Park, J. & Park, A. (2012). Existence, relatedness, or growth? Examining turnover intention of public child welfare caseworkers from a human needs approach. Children and Youth Services Review, 34(10), 2088-2093. https://doi.org/10.1016/j.childyouth.2012.07.002
- [Background] Boyas, J. & Wind, L. H. (2010). Employment-based social capital, job stress, and employee burnout: A public child welfare employee structural model. Children and Youth Services Review, 32(3), 380-388. https://doi.org/10.1016/j.childyouth.2009.10.009
- [Background] Borntrager, C., Caringi, J. C., van den Pol, R., Crosby, L., O'Connell, K., Trautman, A. & McDonald, M. (2012). Secondary traumatic stress in school personnel. Advances in School Mental Health Promotion, 5(1), 38-50. https://doi.org/10.1080/1754730x.2012.664862
- [Background] Sprang G, Craig C, Clark J. Secondary traumatic stress and burnout in child welfare workers: a comparative analysis of occupational distress across professional groups. Child Welfare. 2011;90(6):149-68. PMID 22533047
- [Background] Schaufeli WB, Desart S, De Witte H. Burnout Assessment Tool (BAT)-Development, Validity, and Reliability. Int J Environ Res Public Health. 2020 Dec 18;17(24):9495. doi: 10.3390/ijerph17249495. PMID 33352940
- [Background] Rienks SL. An exploration of child welfare caseworkers' experience of secondary trauma and strategies for coping. Child Abuse Negl. 2020 Dec;110(Pt 3):104355. doi: 10.1016/j.chiabu.2020.104355. Epub 2020 Jan 14. PMID 31948676
- [Background] Prost SG, Middleton JS. Professional quality of life and intent to leave the workforce: Gender disparities in child welfare. Child Abuse Negl. 2020 Dec;110(Pt 3):104535. doi: 10.1016/j.chiabu.2020.104535. Epub 2020 May 22. PMID 32448643
- [Background] Koeske GF, Kelly T. The impact of overinvolvement on burnout and job satisfaction. Am J Orthopsychiatry. 1995 Apr;65(2):282-92. doi: 10.1037/h0079622. PMID 7611345
- [Background] Kliem S, Mossle T, Rehbein F, Hellmann DF, Zenger M, Brahler E. A brief form of the Perceived Social Support Questionnaire (F-SozU) was developed, validated, and standardized. J Clin Epidemiol. 2015 May;68(5):551-62. doi: 10.1016/j.jclinepi.2014.11.003. Epub 2014 Nov 13. PMID 25499982
- [Background] Hannah B, Woolgar M. Secondary trauma and compassion fatigue in foster carers. Clin Child Psychol Psychiatry. 2018 Oct;23(4):629-643. doi: 10.1177/1359104518778327. Epub 2018 May 31. PMID 29848049
- [Background] Dagan SW, Ben-Porat A, Itzhaky H. Child protection workers dealing with child abuse: The contribution of personal, social and organizational resources to secondary traumatization. Child Abuse Negl. 2016 Jan;51:203-11. doi: 10.1016/j.chiabu.2015.10.008. Epub 2015 Nov 6. PMID 26549769
- [Background] Conrad D, Kellar-Guenther Y. Compassion fatigue, burnout, and compassion satisfaction among Colorado child protection workers. Child Abuse Negl. 2006 Oct;30(10):1071-80. doi: 10.1016/j.chiabu.2006.03.009. Epub 2006 Oct 2. PMID 17014908
- [Background] Bridger KM, Binder JF, Kellezi B. Secondary Traumatic Stress in Foster Carers: Risk Factors and Implications for Intervention. J Child Fam Stud. 2020;29(2):482-492. doi: 10.1007/s10826-019-01668-2. Epub 2019 Nov 28. PMID 32431483
- [Background] Adams RE, Boscarino JA, Figley CR. Compassion fatigue and psychological distress among social workers: a validation study. Am J Orthopsychiatry. 2006 Jan;76(1):103-8. doi: 10.1037/0002-9432.76.1.103. PMID 16569133
- See also: Official government page describing the structure and mission of the Flemish integrated youth care system, relevant to the study context. — https://www.jeugdhulp.be/over-jeugdhulp
- See also: Annual public report offering data and background information about Flemish youth care services, providing contextual background for the study. — https://www.jaarverslagjeugdhulp.be
- See also: Official ProQOL site providing validated materials, scoring manuals, and information about the Professional Quality of Life framework. — https://proqol.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT07384026/Prot_SAP_000.pdf